CLINICAL TRIAL: NCT02301728
Title: Short Chain Fatty Acids in Breast Milk
Brief Title: Study on Short Chain Fatty Acids Concentration in Breast Milk and Its Correlation With the Maternal Diet
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Annalisa Passariello, MD, PhD, Federico II University
Other Study IDs: BMB-100
Record Dates: First submitted 2014-11-15; First posted 2014-11-26 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Short Chain Fatty Acids Concentration in Breast Milk
Keywords: breast milk; short chain fatty acids; maternal diet

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Other: sampling of breast milk, obtaining information about the maternal diet — take samples of 3 ml breast milk and 3-days diet diaries

SUMMARY:
The purpose of this study is to determine whether the acetate, butyrate and propionate concentration in breast milk and to evaluate the possible correlation of these concentrations with maternal diet.

ELIGIBILITY:
Inclusion Criteria:

* parturients women at term hospitalized in the Department of Obstetrics, Gynecology and Pathophysiology of Human Reproduction, "Federico II" University of Naples.

Exclusion Criteria:

* infections,
* diabetes and other chronic diseases at the level of each organ or system,
* diseases of pregnancy.
* antibiotics, prebiotics, probiotics and synbiotics in the 30 days prior to the first observation.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: parturients women at term hospitalized in the Department of Obstetrics, Gynecology and Pathophysiology of Human Reproduction, "Federico II" University of Naples.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-01 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
butyrate, acetate and propionate concentration | 10 days after delivery and every 30 days until the fifth month after delivery

SECONDARY OUTCOMES:
Relationship between short chain fatty acids in breast milk and maternal diet (amount of fibers in maternal diet and based on this it will evaluate the variations in short chain fatty acids concentration) | 10 days after delivery and every 30 days until the fifth month after delivery
  Relationship between short chain fatty acids in breast milk and maternal diet will be measured by assessing the amount of fibers in maternal diet and based on this it will evaluate the variations in short chain fatty acids concentration. These assessments will be carried out by using a food diary carefully compiled by mothers before each sampling of breast milk

CONTACTS AND LOCATIONS:
Overall Officials: Annalisa Passariello, MD, PhD, Principal Investigator — "Federico II" University of Naples
Locations (1):
- "Federico II" University of Naples, Naples, Naples, Italy

REFERENCES:
- [Background] Topping DL, Clifton PM. Short-chain fatty acids and human colonic function: roles of resistant starch and nonstarch polysaccharides. Physiol Rev. 2001 Jul;81(3):1031-64. doi: 10.1152/physrev.2001.81.3.1031. PMID 11427691
- [Background] Macfarlane S, Macfarlane GT. Regulation of short-chain fatty acid production. Proc Nutr Soc. 2003 Feb;62(1):67-72. doi: 10.1079/PNS2002207. PMID 12740060
- [Background] Resta-Lenert S, Truong F, Barrett KE, Eckmann L. Inhibition of epithelial chloride secretion by butyrate: role of reduced adenylyl cyclase expression and activity. Am J Physiol Cell Physiol. 2001 Dec;281(6):C1837-49. doi: 10.1152/ajpcell.2001.281.6.C1837. PMID 11698242
- [Background] Roediger WE. Role of anaerobic bacteria in the metabolic welfare of the colonic mucosa in man. Gut. 1980 Sep;21(9):793-8. doi: 10.1136/gut.21.9.793. PMID 7429343
- [Background] Kunzelmann K, Mall M. Electrolyte transport in the mammalian colon: mechanisms and implications for disease. Physiol Rev. 2002 Jan;82(1):245-89. doi: 10.1152/physrev.00026.2001. PMID 11773614
- [Background] Binder HJ, Mehta P. Short-chain fatty acids stimulate active sodium and chloride absorption in vitro in the rat distal colon. Gastroenterology. 1989 Apr;96(4):989-96. doi: 10.1016/0016-5085(89)91614-4. PMID 2925072
- [Background] Boffa LC, Gruss RJ, Allfrey VG. Manifold effects of sodium butyrate on nuclear function. Selective and reversible inhibition of phosphorylation of histones H1 and H2A and impaired methylation of lysine and arginine residues in nuclear protein fractions. J Biol Chem. 1981 Sep 25;256(18):9612-21. PMID 6270094
- [Background] Belderbos ME, Houben ML, van Bleek GM, Schuijff L, van Uden NO, Bloemen-Carlier EM, Kimpen JL, Eijkemans MJ, Rovers M, Bont LJ. Breastfeeding modulates neonatal innate immune responses: a prospective birth cohort study. Pediatr Allergy Immunol. 2012 Feb;23(1):65-74. doi: 10.1111/j.1399-3038.2011.01230.x. Epub 2011 Nov 22. PMID 22103307